CLINICAL TRIAL: NCT06380361
Title: InvestigatioN of a Smart Probe for Lung lEsion Characterization Using Impedance Technology
Acronym: INSPECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sensome (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SEN-ONCO-1
Record Dates: First submitted 2024-03-27; First posted 2024-04-23 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Lung masses; Lung Nodes; Bronchoscopic biopsy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Patient with suspected lung cancer coming to the hospital for bronchoscopic biopsy will be selected for this trial.
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients will be allocated to the same study arm. (Experimental): During the bronchoscopic biopsy procedure, the study device will be entered through the bronchoscope to the level of the lesion. At lesion level, the BioSpy System sensor will make several measurements of the tumors and peripheral lung nodules and masses.
  Interventions: Device: BioSpy System

INTERVENTIONS:
Device: BioSpy System — One arm only - in all eligible study patients, the study device will be used. In patients with suspicion of lung cancer a bronchoscope will be inserted to navigate to the lesion where a biopsy sample will be taken for histology analysis. In the current trial, the device will be used to perform electrophysiological measurements in the lesion during bronchoscopic biopsy procedure.

SUMMARY:
The objective of the study is to evaluate the feasibility of the BioSpy System sensor to differentiate tissues that are encountered during bronchoscopic biopsy of endobronchial tumors and peripheral lung nodules and masses.

DETAILED DESCRIPTION:
Participants in this study require a lung biopsy to confirm if they have a lung tumour. A biopsy is a procedure where a piece of lung tissue is removed for testing. Current biopsy techniques cannot guarantee the exact location of lung tumours, so biopsies can be taken from healthy tissue.

The BioSpy System (BSS) is a device with a probe, which is placed inside a normal biopsy needle. The tip of the probe contains sensors, that will scan the composition of the tissue which is in contact with the sensors.

The INSPECT study aims at collecting the sensor data, with the goal of being able to differentiate the different tissues.

All study participants will have a biopsy with the BSS. Participants will have a hospital visit for the procedure, and will have to stay up to 16 hours after their procedure as per normal hospital practice.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Subjects with lesions eligible for lung biopsy under general anesthesia.
3. Lesion localization:

   1. Central or proximal lesions ≥ 10 mm in diameter confirmed by imaging (CT scan and/or PET scan) and/or endobronchial visual control; or
   2. Peripheral lesions ≥ 20 mm in diameter confirmed by imaging (CT scan and/or PET scan) and/or ultrasound analysis (RP EBUS with central localization of the ultrasound probe) during the procedure.
4. Written Informed Consent to participate in the study.

Exclusion Criteria:

1. Target lesion <10 mm for central and <20 mm for peripheral lesions (as determined on previous imaging)
2. Contra-indication to bronchoscopy procedures
3. Contra-indication to general anesthesia
4. Any subject that is, according to the discretion of the investigator, not eligible for study participation
5. Known lactating or confirmation of positive pregnancy test according to site specific standard of care (e.g. test, verbal communication)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
The ability of BioSpy System to acquire electrophysiological measurements in the relevant tissues during bronchoscopic biopsy. | During the bronchoscopic biopsy procedure
  This endpoint represents the procedural success rate being defined as the BioSpy System obtaining at least one non-anomalous impedance measurement in the lesion during the procedure.

SECONDARY OUTCOMES:
The ability of BioSpy Sysem to differentiate the lesion from healthy tissue | During the bronchoscopic biopsy procedure
  The ability of BioSpy Sysem (BSS) to differentiate the lesion (nodule or mass) from healthy tissue (bronchial tissue, lung parenchyma, …) by means of the impedance measurements.
  These impedance measurements of the BSS will be compared to the physician's assessment based on available imaging (visual control, ultrasound, fluoroscopy etc…) for verification.
  The ability to differentiate tissues will be reported by descriptive statistics.
  To further assess this secondary endpoint, Machine Learning analysis will be applied.
  Following standard procedure, features will be extracted from the impedance measurements and used for model inference.
The ability of BioSpy Sysem to differentiate various lesion types | During the procedure
  The ability of BioSpy Sysem to differentiate various lesion types such as, but not limited to:
  * Tumoral tissue
  * Inflamed tissue
  * Necrotic tissue
  * Fibrosis The impedance measurements of BSS in the lesion will be compared to the histopathology analysis of the collected tissue during the biopsy.
  The ability to differentiate tissues will be reported by descriptive statistics.
  To further assess this secondary endpoint, Machine Learning analysis will be applied.
  Following standard procedure, features will be extracted from the impedance measurements and used for model inference.

CONTACTS AND LOCATIONS:
Locations (2):
- Royal Brisbane and Women's Hospital, Brisbane, Queensland, Australia
- Marie-Lannelongue Hospital, Le Plessis-Robinson, France

IPD SHARING:
Plan to Share IPD: No